CLINICAL TRIAL: NCT04205175
Title: A Single-center, Open-Label, Dose Escalation Study Evaluating the Safety of in Vivo Administration of FEIBA in Congenital Hemophilia A Patients With Inhibitors on Emicizumab
Brief Title: A Study to Evaluate the Safest Dose Range for FEIBA in Hemophilia A Patients With Inhibitors on Emicizumab
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Children's Hospital Los Angeles (Other)
Collaborators: Takeda (Industry)
Responsible Party: Principal Investigator, Guy Young, MD, professor, Children's Hospital Los Angeles
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19 00367
Record Dates: First submitted 2019-12-05; First posted 2019-12-19 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-03

CONDITIONS: Hemophilia A With Inhibitor
MeSH Terms: interventions — anti-inhibitor coagulant complex

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Feiba — This is a single center, open label, dose escalation study of in vivo administration of Feiba in congenital hemophilia A patients with inhibitors who are on emicizumab.

SUMMARY:
Hemophilia A is a severe, life-long, genetic bleeding disorder characterized by a deficiency of factor VIII (FVIII), a crucial cofactor of the coagulation system. The mainstay of hemophilia treatment is factor replacement therapy with FVIII clotting factor concentrates (CFC) and these can be given episodically in response to bleeding or prophylactically to prevent bleeding. The main adverse effect of FVIII CFC is the development of neutralizing anti-drug antibodies termed inhibitors, and these render replacement therapy less effective if they are low titer inhibitors or completely ineffective if they are of the high titer variety. These so-called 'inhibitor patients' cannot rely on FVIII CFC for their treatment and are treated with other CFC called bypassing agents such as activated prothrombin complex concentrate (aPCC/Feiba). While these agents can be effective in some patients for prophylaxis, they are not as effective for bleed prevention as FVIII CFC for patients without inhibitors.Recently, emicizumab (Hemlibra, Roche), was developed and licensed for the prevention of bleeding in patients with hemophilia A with and without inhibitors. However, patients in the clinical trials for emicizumab have developed thrombotic adverse events and only patients who received doses of Feiba of >100 IU/kg/24 hours for more than 24 hours developed thrombosis.

As a result of the above data, recommendations have been to either avoid altogether in patients on emicizumab, or to be very cautious about using it to treat breakthrough bleeding. With this in mind, we propose to study the in vivo combination of Feiba in patients with inhibitors on emicizumab.

DETAILED DESCRIPTION:
Explanation of the study: Hemophilia A is a severe, life-long, genetic bleeding disorder characterized by a deficiency of factor VIII (FVIII), a crucial cofactor of the coagulation system. The mainstay of hemophilia treatment is factor replacement therapy with FVIII clotting factor concentrates (CFC) and these can be given episodically in response to bleeding or prophylactically to prevent bleeding. The main adverse effect of FVIII CFC is the development of neutralizing anti-drug antibodies termed inhibitors, and these render replacement therapy less effective if they are low titer inhibitors or completely ineffective if they are of the high titer variety. These so-called 'inhibitor patients' cannot rely on FVIII CFC for their treatment and are treated with other CFC called bypassing agents such as activated prothrombin complex concentrate (aPCC/Feiba). While these agents can be effective in some patients for prophylaxis, they are not as effective for bleed prevention as FVIII CFC for patients without inhibitors.Recently, emicizumab (Hemlibra, Roche), was developed and licensed for the prevention of bleeding in patients with hemophilia A with and without inhibitors. However, patients in the clinical trials for emicizumab have developed thrombotic adverse events and only patients who received doses of Feiba of >100 IU/kg/24 hours for more than 24 hours developed thrombosis.

Rationale: As a result of the above data, recommendations have been to either avoid altogether in patients on emicizumab, or to be very cautious about using it to treat breakthrough bleeding. With this in mind, we propose to study the in vivo combination of Feiba in patients with inhibitors on emicizumab.

Intervention: Administration of Feiba on the lower end of the licensed doses (or lower) and running thrombin generation assay (TGA) in patients on emicizumab.

Objectives: To demonstrate the thrombin generation of the in vivo administration of Feiba at various doses to patients with congenital hemophilia A and inhibitors who are on emicizumab and to assess the safety of a single Feiba infusion in patients with congenital hemophilia A with inhibitors.

Study population: Male patients with congenital hemophilia A of any severity and any age with a history of high titer factor VIII inhibitor who are currently treated with emicizumab for a minimum of 2 months without interruption.

Study methodology: Patients who agree to participate will be infused a single, weight-based dose at each visit in the Infusion Center or the Outpatient Clinic. Depending on the thrombin generation of each individual patient following the initial dose, the study team will schedule the next infusion visit for subsequent Feiba dose.

Study endpoint: Once any patient on this trial achieves normal or near normal (within 10%) thrombin generation, they will not receive subsequent Feiba infusions even if that occurs after the lowest dose. Thus, no patient is expected to have excessive thrombin generation.

Statistics: The study will only employ descriptive statistics. The main outcome measure will be to determine the dose of Feiba that most closely approximates normal thrombin generation in patients with congenital hemophilia A with inhibitors who are on emicizumab.

Plans for analysis: the goal is to complete all study procedures within 12 months and have 2 months for data analysis and evaluation. Overall the goal is to complete the project including a submission for an abstract and publication within 14 months from the start of patient accrual.

ELIGIBILITY:
Inclusion Criteria:

1. Male patients with congenital hemophilia A of any severity and any age.
2. History of high titer factor VIII inhibitor (Bethesda unit >5)
3. Currently prescribed bypassing agent therapy for bleed management.
4. Current treatment with emicizumab for a minimum of 2 months without interruption.

Exclusion Criteria:

1. Active bleed requiring factor therapy at screening.
2. Treatment with rFVIIa or aPCC 7 days prior to screening.
3. Surgical procedure 14 days prior to screening.
4. Current use of any medication other than emicizumab that could affect the coagulation system e.g. aspirin, anticoagulants, etc.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Since Hemophilia is a X-linked bleeding disorder occurring mostly in males we expected to mostly enroll male-identified subjects.
Enrollment: 20 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Thrombin generation | The goal is to complete all study procedures within 12 months.
  Thrombin generation capacity of the patients will be measured after every Feiba infusion with Thrombin Generation Assay.

CONTACTS AND LOCATIONS:
Overall Officials: Guy Young, MD, Principal Investigator — professor
Locations (1):
- Childrens Hospital Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes